CLINICAL TRIAL: NCT05875519
Title: Evaluation of Healing Process and Blood Sugar Level Following Local Anesthetic Infiltration With and Without Vasoconstrictor for Extraction of Maxillary Teeth in Diabetic Patients Double Blind Randomized Clinical Trial
Brief Title: Healing Process and Blood Sugar Level Following Local Anesthetic Infiltration With and Without Vasoconstrictor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 714
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-05

CONDITIONS: Diabetes; Anesthesia, Local
MeSH Terms: conditions — Diabetes Mellitus | interventions — Anesthesia, Local; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaesthesia with vasocontrictor (Experimental)
  Interventions: Drug: Local anaesthesia with vasocontrictor (Mepivacaine hydrochloride 20 mg (2%) + Levonordefrin hydrochloride 0.06 mg)
- Anaesthesia without vasocontrictor (Active Comparator)
  Interventions: Drug: Local anaesthesia with vasocontrictor (Mepivacaine hydrochloride 20 mg (2%) + Levonordefrin hydrochloride 0.06 mg)

INTERVENTIONS:
Drug: Local anaesthesia with vasocontrictor (Mepivacaine hydrochloride 20 mg (2%) + Levonordefrin hydrochloride 0.06 mg) — Mepivacaine hydrochloride 20 mg (2%) + Levonordefrin hydrochloride 0.06 mg

SUMMARY:
Evaluating the healing of the extraction socket and the glycemic levels before, and after injection of local anesthesia with and without vasoconstrictor in diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria patients over 20 years and under 60 years of age
* DM controlled by medication
* Requiring a tooth extraction in the maxilla, with an indication of the intra-alveolar technique for periodontal reasons.
* Only participants that are willing to control and record blood glucose level throughout the study period.

Exclusion Criteria:

* Patients with any significant medical condition (besides DM)
* Alcoholic individuals
* Patients on drugs that affect the central nervous systems
* Patients who reported the use of drugs that might interfere with pain sensitivity
* Pregnant and lactating women
* Patients with hypersensitivity to local anesthetics or non-steroidal anti-inflammatory drugs (NSAIDs).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Glycemic level recorded before local anesthesia administration and 30 minutes following local anesthesia injection using glucometer | 30 minutes

SECONDARY OUTCOMES:
Healing score of the extraction socket | 21 days
  4 = Necrotic Tissue (Eschar): black, brown, or tan tissue that adheres firmly to the wound bed 3 = Slough: yellow or white tissue that adheres to the wound bed 2 = Granulation Tissue: pink or beefy red tissue with a shiny, moist, granular appearance.
  1 = Epithelial Tissue: for superficial ulcers, new pink or shiny tissue that grows in from the edges or as islands on the wound surface.
  0 = Closed/Resurfaced: the wound is completely covered with epithelium.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided